FWA 00032748 July 4, 2024

IORG0011243

## Management of Postspinal Anesthesia Hypotension Duing Elective Cesarean Section: Baby Norepinephrine Versus Ephedrine

## **Consent Form for Participation in Clinical Research**

**Research title:** Management of Postspinal Anesthesia Hypotension During Elective Cesarean Section: Baby Norepinephrine Versus Ephedrine

The objectives and modalities of the study about « Management of Postspinal Anesthesia Hypotension During Elective Cesarean Section: Baby Norepinephrine Versus Ephedrine » were clearly explained to me by Dr HAFYENE ABDELMAJID. I have read and understood the information sheet that was given to me. I agree that the documents in my medical file that relate to the study may be accessible to the study leaders and health authorities.

With the exception of these people, who will process the information in the strictest respect of medical confidentiality, my anonymity will be preserved.

I understand that my participation in the study is voluntary. I am free to refuse to participate and I am free to withdrawfrom the research at any time. My refusal to participate or withdrawal of concent will not affect the quality of care I will receive in any way. My consent does not relieve the organizers of this study of their responsibilities. I retain all my rights guaranteed by law.

After discussing it and having obtained the answers to all my questions, I freely and voluntarily agree to participate in this research.

| Participant's Name and Signature: |
|-----------------------------------|
| Date : |
| nvestigator's signature: |
| Date : |